CLINICAL TRIAL: NCT01221766
Title: The Impact of Adnexal Involvement of the Severity and Prognosis of Chronic Graft-versus-Host Disease
Brief Title: Impact of Adnexal Involvement of the Severity and Prognosis of Chronic Graft-versus-Host Disease
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Huang, MD, Instructor in Dermatology, Dana-Farber Cancer Institute
Other Study IDs: 10-163
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Graft vs Host Disease; Chronic Graft vs Host Disease; cGVHD
Keywords: adnexal; hair and nail; chronic graft vs host disease; children
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This research study will help us learn more about how chronic graft-versus-host disease affects the skin, hair and nails. We are interested in knowing if hair and nail problems predict worse disease. This information may help us treat patients like you in the future.

DETAILED DESCRIPTION:
* At the initial visit, participants will have a complete examination of their skin, hair and nails. We will also test muscle strength and movement by moving the participant's arms, legs and neck. Photographs will be taken of the skin, hair and nails of they are abnormal. Blood tests will be done to check the liver and blood cell count. The participant and their legal guardian will answer questions about how the participant feels and about their health.
* Participants will then be scheduled for follow up visits at 3 months, 6 months, and 12 months. At each subsequent visit the following will be done: A complete examination of the skin, hair and nails; a test of muscle strength; photographs will be repeated; blood tests to check liver and blood cell counts; and questions about how the participant feels and about their health.

ELIGIBILITY:
Inclusion Criteria:

* Received hematopoietic stem cell transplant
* Meet the diagnostic criteria for cutaneous cGVHD

Exclusion Criteria:

* Previous HSCT (other then the current HSCT)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research subject population is children who have received hematopoietic stem cell transplant and developed chronic graft-versus-host disease. All children seen at the pediatric GVHD clinic at the Dana-Farber Cancer Institute will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Adnexal involvement | 1 year
  To determine if adnexal involvement predicts worse severity and/or prognosis in chronic GVHD. This will be measured by administration of systemic therapy other than steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huang, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts